CLINICAL TRIAL: NCT05689671
Title: Atezolizumab/Carboplatin/Nab-Paclitaxel vs. Pembrolizumab/Platinum/Pemetrexed in Metastatic TTF-1 Negative Lung Adenocarcinoma
Brief Title: Pemetrexed-free vs. Pemetrexed-based Immunochemotherapy in Metastatic TTF-1 Negative Lung Adenocarcinoma
Acronym: ANTELOPE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nikolaj Frost MD (Other)
Collaborators: Roche Pharma AG (Industry); Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor-Investigator, Nikolaj Frost MD, Nikolaj Frost, PD Dr. med., Principal Investigator, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAP131705; 2022-002990-27 (EudraCT Number); AIO-TRK-0122 (Other: Arbeitsgemeinschaft Internistische Onkologie)
Record Dates: First submitted 2022-11-30; First posted 2023-01-19 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer Metastatic
Keywords: NSCLC; checkpoint inhibitors; immunochemotherapy
MeSH Terms: interventions — atezolizumab; Taxes; Albumin-Bound Paclitaxel; Carboplatin; pembrolizumab; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pemetrexed-free Immunochemotherapy (Arm A) (Experimental): Atezolizumab 1200 mg q3w, carboplatin AUC 5-6 q3w, nab-paclitaxel 100 mg/m2 qw (administered for 4 cycles with subsequent maintenance with atezolizumab monotherapy 1200 mg q3w until loss of clinical benefit or occurrence of unacceptable toxicity)
  Interventions: Drug: Atezolizumab; Drug: Nab paclitaxel; Drug: Carboplatin
- Pemetrexed-based Immunochemotherapy (Arm B) (Active Comparator): Pembrolizumab 200 mg q3w, cisplatin 75 mg/m2 q3w OR carboplatin AUC 5-6 (each) q3w, pemetrexed 500 mg/m2 q3w (administered for 4 cycles with subsequent maintenance with pembrolizumab 200 mg AND pemetrexed 500 mg/m2 (each) q3w until loss of clinical benefit or occurrence of unacceptable toxicity)
  Interventions: Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Atezolizumab — 1200 mg i.v. q3w
  Other Names: Tecentriq
  Arms: Pemetrexed-free Immunochemotherapy (Arm A)
Drug: Nab paclitaxel — 100 mg/m² i.v. qw
  Other Names: Abraxane
  Arms: Pemetrexed-free Immunochemotherapy (Arm A)
Drug: Carboplatin — AUC 5-6 i.v. q3w
  Arms: Pemetrexed-free Immunochemotherapy (Arm A)
Drug: Pembrolizumab — 200 mg i.v. q3w
  Other Names: Keytruda
  Arms: Pemetrexed-based Immunochemotherapy (Arm B)
Drug: Cisplatin — 75 mg/m² i.v. q3w
  Arms: Pemetrexed-based Immunochemotherapy (Arm B)
Drug: Carboplatin — AUC 5-6 i.v. q3w
  Arms: Pemetrexed-based Immunochemotherapy (Arm B)
Drug: Pemetrexed — 500 mg/m² i.v. q3w
  Arms: Pemetrexed-based Immunochemotherapy (Arm B)

SUMMARY:
This is an open-label randomized, controlled, multicenter, phase II trial with two arms. Patients with metastatic TTF-1 negative, treatment-naive lung adenocarcinoma without actionable genomic alterations are randomized in a 1:1 manner to investigate the efficiency of atezolizumab, carboplatin and nab-paclitaxel (Arm A) versus pembrolizumab, cis-/carboplatin and pemetrexed (Arm B) as first-line treatment.

DETAILED DESCRIPTION:
Thyroid transcription factor 1 (TTF-1) is expressed in the majority of lung adenocarcinoma and has a clear prognostic value. Pemetrexed-based immunochemotherapy is a standard of care for advanced lung adenocarcinoma. However, real-world data suggest that TTF-1 negative patients might derive superior outcome using pemetrexed-free regimens. The aim of this study is to compare a pemetrexed-free (Arm A) vs. a pemetrexed-based immunochemotherapy (Arm B) as first-line treatment for metastatic TTF-1 negative lung adenocarcinoma without actionable genomic alterations.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided written informed consent
2. Patient* 18 years or older at time of signing the informed consent form
3. Histologically or cytologically confirmed metastatic stage IV non-squamous NSCLC
4. Negative local testing for TTF-1
5. Negative molecular testing for EGFR mutations and ALK rearrangements (tested locally). Exception: In specific individual cases, treatment can be initiated prior to receiving molecular diagnostics after consulting with the sponsor, if the local principal investigator assesses the likelihood of an EGFR mutation or ALK fusion to be negligible. However, this should only be done in exceptional cases if the patient has particularly high demand for treatment. If it is subsequently found that patients are positive for EGFR mutations and/or ALK rearrangements, they must be withdrawn from the study immediately and must not receive any further study medication. Instead, patients should receive adequate SOC therapy outside the study.

   Awaiting results for molecular testing remains standard procedure for patient inclusion.
6. PD-L1 tumor proportion score (TPS) < 50%, tested locally by QUiP®-certified immunohistochemistry
7. ECOG performance status ≤ 1
8. Measurable lesions according to RECIST v1.1
9. Life expectancy ≥ 12 weeks
10. Adequate hepatic, renal and bone marrow function

    1. Hemoglobin ≥ 8.0 g/dL
    2. Absolute neutrophil count ≥ 1.5 x 109/L
    3. Platelets ≥ 100 x 109/L
    4. Calculated creatine clearance ≥ 50 mL/min as determined by the Cockcroft-Gault equation and/or creatinin ≤ 1,5x upper limit of normal (ULN)
    5. Serum bilirubin ≤ 1.5 x institutional ULN
    6. AST/ ALT and alkaline phosphatase ≤ 2.5 x ULN
    7. International normalized ratio (INR)/ Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PTT is within therapeutic range of intended use of anticoagulants
11. The patient is willing and able to comply with the protocol for the duration of the study, including hospital visits for treatment and scheduled follow-up visits and examinations.
12. Female patients who are considered as woman of childbearing potential (WOCBP) must use any contraceptive method with a failure rate of less than 1% per year during the treatment as well as up to 6 months after the last dose of study treatment. Male patients who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year during the treatment as well as at least 6 months after the last dose of IMP. Female patients who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) as well as azoospermic male patients do not require contraception

Exclusion Criteria:

1. Mixed histologies (small-cell and non-small cell or non-squamous and squamous; patients exhibiting the latter expression pattern may be eligible if the non-squamous part predominates)
2. Patients having received:

   1. Systemic treatment for metastatic or locally advanced disease
   2. prior PD-1/PD-L1 immunotherapies (prior treatment with CD137 agonists or immune checkpoint blockade therapies, including, but not limited to, anti-cytotoxic T lymphocyte associated protein 4 [anti-CTLA-4], anti T cell immunoreceptor with Ig and tyrosine-based inhibition motif domains [anti-TIGIT], anti-PD-1 and anti-PD-L1 therapeutic antibodies)
3. Symptomatic, neurologically unstable CNS metastases or requiring increasing doses of steroids to manage CNS symptoms within 2 weeks prior to study entry (maximal acceptable dose must be ≤ 10 mg of prednisolone). Patients with asymptomatic, incidentally detected CNS metastases may be enrolled. Palliative radiotherapy for asymptomatic brain metastases (and any other, non-brain metastases, e.g. bone metastases) may be conducted after study entry.
4. Leptomeningeal disease
5. History of interstitial lung disease
6. Severe infection within 2 weeks prior to study entry. Clinical signs must have been resolved to CTCAE grade ≤ 1
7. Active infection with hepatitis B or C virus (HBV, HCV), human immunodeficiency virus (HIV) or Mycobacterium tuberculosis
8. Known additional malignancies other than NSCLC, either untreated or having required active treatment within the past 3 years
9. Significant cardiovascular disease (≥ NYHA 3)
10. Active or prior documented autoimmune or inflammatory disorders (including but not limited to diverticulitis [with the exception of diverticulosis], celiac disease, systemic lupus erythematosus, Sarcoidosis, or Wegener's syndrome [granulomatosis with polyangiitis], Graves' disease, rheumatoid arthritis, hypophysitis, uveitis). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (e.g., following Hashimoto's disease) stable on hormone replacement
    3. Patients with controlled Type I diabetes mellitus on an insulin regimen
    4. Any chronic skin condition that does not require systemic therapy
    5. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
11. Current or prior use of immunosuppressive medication within 14 days before the first dose of atezolizumab/pembrolizumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g. intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication)
12. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and IL-2) within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment
13. Live vaccine within 30 days prior to first dose of trial treatment
14. Known allergy or hypersensitivity to any component of the chemotherapy regimen or to atezolizumab or pembrolizumab or any constituents of the products
15. Any co-existing medical condition that in the investigator's judgement will substantially increase the risk associated with the patient's participation in the study.
16. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 30 months
  time from randomization to the date of death due to any case

SECONDARY OUTCOMES:
Objectice Response Rate (ORR) | 30 months
  proportion of subjects with best response of complete or partial response (CR & PR) according to RECIST v1.1
Progression-Free Survival (PFS) | 30 months
  time from randomization until progression defined by RECIST v1.1 or death due to any cause
One-Year Overall Survival Rate | 30 months
  percentage of patients alive at 12 months after randomization
Time to Next Treatment or Death (TNTD) | 30 months
  time from initial study randomization to the start of next subsequent treatment or death, whichever occurs first
Progression-Free Survival 2 (PFS2) | 30 months
  time from initial study randomization to second disease progression or death from any cause to assess efficacy post-trial-treatment anti-cancer therapy
Health-related quality of life 1 (HRQoL) | Assessed after randomization at cycle 1 day 1, after completion of cycle 4 (each cycle is 21 days) of the chemoimmunotherapy and at progressive disease (if occurring within the maximum time frame of 30 months)
  assessed with the QoL questionnaire QLQ-C30 on general health conditions in lung cancer patients using numeric scales ranging from 1-4. Lower numbers indicate no, higher numbers high agreement.
Health-related quality of life 2 (HRQoL) | Assessed after randomization at cycle 1 day 1, after completion of cycle 4 (each cycle is 21 days) of the chemoimmunotherapy and at progressive disease (if occurring within the maximum time frame of 30 months)
  assessed with the lung cancer symptom-specific QoL questionnaire QLQ-LC13 using numeric scales ranging from 1-4. Lower numbers indicate no, higher numbers high agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaj Frost, PD Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (36):
- Germany (36):
  - Klinikum St. Marien, Amberg
  - Universitätsklinikum Augsburg, Augsburg
  - MVZ Taunus GmbH, Bad Homburg
  - Evangelische Lungenklinik Krankenhausbetriebs gGmbH, Berlin
  - Evangelische Lungenklinik, Berlin
  - Charité Universitätsmedizin, Berlin
  - Helios Klinikum Emil von Behring, Berlin
  - Klinikum Bielefeld, Bielefeld
  - Kliniken der Stadt Köln GmbH, Cologne
  - Technische Universität Dresden Medizinische Fakultät Carl Gustav Carus, Dresden
  - Universitätsklinikum Essen, Essen
  - KEM Evang. Kliniken Essen-Mitte, Essen
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Krankenhaus Nordwest, Frankfurt
  - Universitätsklinikum Frankfurt am Main, Frankfurt am Main
  - Asklepios Klinik Gauting GmbH, Gauting
  - Universitätsmedizin Göttingen, Göttingen
  - LungenClinic Großhansdorf GmbH, Großhansdorf
  - Asklepios Klinkum Hamburg, Hamburg
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Thoraxzentrum Ruhrgebiet Ev. Krankenhaus Herne, Herne
  - Helios Klinikum Krefeld, Krefeld
  - ÜBAG- Medizinisches Versorgungszentrum Dr. Vehling-Kaiser GmbH, Landshut
  - Klinikum Lippe GmbH, Lemgo
  - Klinikum Ludwigsburg, Ludwigsburg
  - UKSH, Campus Lübeck, Lübeck
  - Medizinische Fakultät Mannheim der Universität Heidelberg, Mannheim
  - LMU Klinikum, München
  - Unversitätsklinikum Münster, Münster
  - Überörtliche Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Pius Hospital, Oldenburg
  - MVZ für Hämatologie und Onkologie Ravensburg GmbH, Ravensburg
  - Barmherzige Brüder Krankenhaus Regensburg, Regensburg
  - Elblandkliniken Stiftung & Co. KG Elblandklinikum Riesa, Riesa
  - Klinikum Stuttgart, Stuttgart

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frost N, Zhamurashvili T, von Laffert M, Klauschen F, Ruwwe-Glosenkamp C, Raspe M, Brunn M, Ochsenreither S, Temmesfeld-Wollbruck B, Suttorp N, Grohe C, Witzenrath M. Pemetrexed-Based Chemotherapy Is Inferior to Pemetrexed-Free Regimens in Thyroid Transcription Factor 1 (TTF-1)-Negative, EGFR/ALK-Negative Lung Adenocarcinoma: A Propensity Score Matched Pairs Analysis. Clin Lung Cancer. 2020 Nov;21(6):e607-e621. doi: 10.1016/j.cllc.2020.05.014. Epub 2020 May 22. PMID 32620471
- See also: Study description on the webpage of the "Oncology in Internal Medicine Working Group" (AIO) within the German Cancer Society — https://www.aio-portal.de/studie/176--antelope.html